CLINICAL TRIAL: NCT07404839
Title: Scaling up Building Healthy Families in Rural Areas and Small Towns
Brief Title: Scaling up Building Healthy Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennie Hill, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00188809; R01DK142843 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity, Child
Keywords: rural; implementation strategies; family based program; dissemination and implementation science; lifestyle change intervention; family based programs
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Hybrid type three effectiveness-implementation community-level randomized control trial in which communities will be recruited and assigned to one of two study conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Building Healthy Families (BHF) Program Resources Package Only (BHF-PO) (Active Comparator): The BHF Program Resources include an online train-the-trainer system, program materials, and a data portal for use by community-based implementation teams. Communities randomized to the BHF Program Resources Package Only (BHF-PO) study condition will have access to the online train-the-trainer system, program materials, and a data portal for use by community-based implementation teams. Community-based implementation teams (CITs) will use the BHF Program Resources to train and deliver the BHF Program to families in their community.
  Interventions: Behavioral: Building Healthy Families Program
- Building Healthy Families Learning Collaborative (BHF-LC). (Experimental): Communities randomized to the BHF-LC study condition have access to BHF Program Resources and enhanced training through the learning collaborative facilitation strategy. Community Implementation Team (CIT) members in this study condition will participate in the learning collaborative, which consists of quarterly virtual learning sessions (8 total), over a two-year period. In between learning sessions, each BHF-LC CIT will have a 1-hour 1:1 action period meeting with the research team.
  Community-based implementation teams (CITs) will use the BHF Program Resources to train and deliver the BHF Program to families in their community.
  Interventions: Behavioral: Building Healthy Families Program

INTERVENTIONS:
Behavioral: Building Healthy Families Program — Building Healthy Families (BHF) is an evidence-based, family-based weight management program designed for children aged 5-13 who are overweight or obese and their parents or caregivers. Family-based weight management programs focus on creating a supportive, positive environment for lifestyle behavior change that promotes healthy growth and development. BHF is a group-based program, and education sessions focus on healthy eating, physical activity, and lifestyle modification for the entire family. The BHF Program consists of 12 weekly education sessions (~2 hours each) and 6 relapse-prevention refresher sessions over 1 year (12 months total). The BHF program meets the current recommendations for intensive health behavior and lifestyle treatment (IHBLT) programs from professional groups, and BHF is a recommended program for community adoption and implementation.
  Other Names: BHF Program

SUMMARY:
Evidence-based interventions for childhood obesity (EBI-CO) can reduce child weight status, but for families living in rural areas and small cities, the availability of interdisciplinary healthcare teams recommended to deliver EBI-CO is low. To address this issue, we adapted an EBI-CO, called Building Healthy Families (BHF), that includes all the materials and training resources necessary for rural program implementation and found, in a pilot study, that when paired with opportunities to learn from the program developers and other community implementation teams packaged program led to effective program delivery across 4 rural communities. In this study, we will scale up our pilot and compare our packaged BHF Resources with and without a learning collaborative facilitation strategy, examining outcomes such as reach, effectiveness, implementation, and potential for sustainability in rural areas.

DETAILED DESCRIPTION:
We propose a community-level randomized control trial to determine the relative utility of providing an online training and resource package to support planning, implementation, and sustainability of an evidence-based childhood obesity treatment intervention (EBI-CO) with and without participation in a systems-based action learning collaborative to improve reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) in rural areas, small towns or other low-resourced communities.

20% of the U.S. population resides in micropolitan (cities <50,000) and rural settings with lower access to preventive health services and behavioral programs to address obesity. While EBI-COs exist, few have been translated into micropolitan and rural settings. A related issue is the potential mismatch between the resources and expertise used to deliver research and hospital-based EBI-COs in urban areas and those in micropolitan and rural areas. To address these issues, we piloted the development and implementation of the Building Healthy Families (BHF) Online Training Resources and Program Package (BHF Program Resources) and implementation blueprint to address childhood obesity in micropolitan and rural areas. The BHF Program Resources include an online train-the-trainer system, program materials, and a data portal for use by community-based implementation teams.

In our pilot study we found that (1) a bundled fund and contract and network weaving strategy to increase BHF adoption was successful at recruiting micropolitan communities to deliver BHF, (2) a systems-based learning collaborative (BHF-LC) implementation strategy was feasible and demonstrated the potential for superior implementation fidelity, and sustainability when compared to receiving the BHF Resources Package Only (BHF-PO), (3) community implementation teams that participated in the BHF-LC reported more positive perceptions of contextual factors, facilitation, and characteristics of BHF when compared to those that did not, and (4) community implementation teams needed additional support related to program reach.

We propose to expand our pilot into a fully powered hybrid Type 3 effectiveness-implementation, community-level RCT to test the utility of BHF-LC to improve BHF reach, effectiveness, implementation, and maintenance when compared to communities that receive the BHF Resources Package Only (BHF-PO). We will scale up our bundled adoption strategy to engage 30 micropolitan and rural communities. We will initiate community recruitment across the 6-state region served by the Huntsman Cancer Institute (Idaho, Montana, Nevada, New Mexico, Wyoming, Utah; See Letters of Support) and expand to rural, frontier, and other low-resourced settings in all states as needed. We will randomly assign communities to either the BHF-PO (n=15) or in combination with the BHF-LC (n=15) to achieve the following aims:

Specific Aim 1: Determine if community implementation teams (a) deliver BHF with higher implementation fidelity (primary outcome), (b) achieve higher reach, and (c) have an increased likelihood of sustainability, based on assignment to BHF-PO or BHF-LC.

Specific Aim 2: Determine the effectiveness of BHF in reducing and maintaining child weight status based on community assignment to BHF-LC versus BHF-PO.

Specific Aim 3: Conduct a cost evaluation and cost-effectiveness analysis comparing communities that participate in the BHF-LC to those that receive the BHF Program Resources (BHF-PO) alone.

ELIGIBILITY:
Communities eligible to participate include those in rural areas or other low-resource settings.

Eligible communities must respond to a call for proposals by submitting a letter of intent and a brief narrative about the local need for BHF and readiness for implementation.

The community is willing to be randomized to either study condition.

The community is willing to create a Community Implementation Team (CIT) to implement BHF.

Community Implementation Teams (CIT) include adults aged 18 and above working at community-based organizations that applied and were selected through the bundled adoption strategy (i.e., LOI/RFA) process.

Families eligible for the BHF Program must have at least one child between the ages of 5 and 13 years with a BMI >85th percentile. One parent or caregiver must agree to attend sessions with the child.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Implementation Fidelity (community level) | From BHF session initiation to the end of sessions (~ 12 months) for one cohort in each enrolled community.
  The primary implementation-fidelity outcome will be measured by direct observation and is defined as the number of session activities completed by the number of sessions delivered.

SECONDARY OUTCOMES:
Change in child weight status | 3 months
  Child participant height, weight, age, and gender data recorded by CITs at baseline and 3 months will be used to calculate the change in weight status (i.e., BMI z-score).
Costs | Up to 24 months
  The cost of program adoption and implementation for communities will be tracked over the study using time-tracking methods to capture the time spent on program activities by implementation staff.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Hill, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified raw and scored summary datasets for the primary outcome (implementation fidelity by site) and secondary outcome (effectiveness-child weight status) will be created for data analysis. Codebooks, programming code for data cleaning and storage, and preliminary and final output tables created during the analysis will also be stored.
  Family-level data from the BHF Resources are accessible only to the study team, and raw data or data with potential family or child-level identifiers cannot be shared. Deidentified summary data may be shared after all potentially revealing information is removed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Deidentified scored datasets for the primary outcome (implementation fidelity by site) will be available at the time of peer review publication and will be available open access for seven years following the end of the trial period.